CLINICAL TRIAL: NCT02116777
Title: A Phase 1/2 Study of BMN 673, an Oral Poly(ADP-Ribose) Polymerase Inhibitor, Plus Temozolomide in Children With Refractory or Recurrent Malignancies
Brief Title: Talazoparib and Temozolomide in Treating Younger Patients With Refractory or Recurrent Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-00804; NCI-2014-00804 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ADVL1411 (Other: Pediatric Early Phase Clinical Trial Network); ADVL1411 (Other: CTEP); UM1CA097452 (NIH)
Record Dates: First submitted 2014-04-15; First posted 2014-04-17 (Estimated); Results first posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Adult Solid Neoplasm; Childhood Solid Neoplasm; Recurrent Childhood Central Nervous System Neoplasm; Recurrent Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Recurrent Malignant Solid Neoplasm; Refractory Central Nervous System Neoplasm
MeSH Terms: conditions — Central Nervous System Neoplasms; Neuroectodermal Tumors, Primitive, Peripheral | interventions — talazoparib; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (talazoparib, temozolomide): Phase 1 (Experimental): (Part A): Patients receive talazoparib PO QD or BID on days 1-6 and temozolomide PO QD on days 2-6. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Talazoparib; Drug: Temozolomide
- Treatment (talazoparib, temozolomide): Phase 2 (Experimental): (Part B): Relapse/Refractory EWS or PNET Patients receive MTD from Phase 1 portion of study. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Talazoparib; Drug: Temozolomide

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Talazoparib — Given PO
  Other Names: BMN 673; BMN-673
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac; TMZ

SUMMARY:
This phase I/II trial studies the side effects and best dose of talazoparib and temozolomide and to see how well they work in treating younger patients with tumors that have not responded to previous treatment (refractory) or have come back (recurrent). Talazoparib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving talazoparib together with temozolomide may work better in treating younger patients with refractory or recurrent malignancies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) of temozolomide when combined with a dose of talazoparib (BMN 673) given once daily for 5 days after a one day dose of BMN 673 administered orally (either once daily or twice daily), every 28 days to children with refractory or recurrent solid tumors. (Phase I) II. To define and describe the toxicities of BMN 673 given with temozolomide administered on this schedule. (Phase I) III. To characterize the pharmacokinetics of BMN 673 and temozolomide when given in combination to children with refractory or recurrent cancer. (Phase I) IV. To define the antitumor activity of BMN 673 when given with temozolomide in recurrent/refractory Ewing sarcoma.(Phase II)

SECONDARY OBJECTIVES:

I. To preliminarily define the antitumor activity of BMN 673 and temozolomide in pediatric patients with recurrent or refractory solid tumors within the confines of a phase I study.

II. To explore possible predictive biomarkers in archival tumor tissue from Ewing sarcoma patients in Phase II.

OUTLINE: This is a phase I, dose-escalation study followed by a phase II study.

Patients receive talazoparib orally (PO) once daily (QD) or twice daily (BID) on days 1-6 and temozolomide PO QD on days 2-6. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Age:

  * Phase 1 (Part A)

    * Patients must be > than 12 months and =< 21 years of age at the time of study enrollment
  * Phase 2 (Part B)

    * Patients must be > than 12 months and =< 30 years of age at the time of study enrollment
* Body surface area (for Parts A and B):

  * Patients must have a body surface area (BSA) of >= 0.42 m^2 at the time of study enrollment
* Diagnosis:

  * Phase 1 (Part A)

    * Solid tumors (Part A1): patients with relapsed or refractory solid tumors including central nervous system (CNS) tumors without bone marrow involvement are eligible; patients must have had histologic verification of malignancy at original diagnosis or relapse except in patients with intrinsic brain stem tumors, optic pathway gliomas, or patients with pineal tumors and elevations of cerebrospinal fluid (CSF) or serum tumor markers including alpha-fetoprotein or beta-human chorionic gonadotropin (HCG)
    * Ewing sarcoma or peripheral primitive neuroectodermal tumor (PNET) (Part A2): patients with relapsed or refractory Ewing sarcoma or peripheral PNET without bone marrow involvement will be eligible for Part A2 if there are no available slots on Part A1; these patients will be enrolled at one dose level below the dose level at which patients on Part A1 are actively enrolling, or at the starting dose level (dose level 1) if dose escalation has not yet occurred; patients must have had histologic verification of malignancy at original diagnosis or relapse
  * Phase 2 (Part B)

    * Ewing sarcoma or peripheral PNET: patients with relapsed or refractory Ewing sarcoma or peripheral PNET are eligible; patients must have had histologic verification of malignancy at original diagnosis or relapse
  * Phase 2 (Part C)
* Disease status:

  * Phase 1 (Part A):

    * Patients must have either measurable or evaluable disease
  * Phase 2 (Part B):

    * Ewing sarcoma or peripheral PNET: patients must have measurable disease
* Therapeutic options: patient's current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life
* Karnofsky >= 50% for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age; Note: neurologic deficits in patients with CNS tumors must have been relatively stable for at least 7 days prior to study enrollment; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients who have received prior therapy with a temozolomide-based regimen are eligible; Note: patients who have progressed on a poly adenosine diphosphate ribose polymerase (PARP) inhibitor and temozolomide regimen are not eligible for Part A of the study
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer chemotherapy

  * Myelosuppressive chemotherapy:

    * Solid tumors (Part A and Part B): at least 21 days after the last dose of myelosuppressive chemotherapy (42 days if prior nitrosourea)
  * Hematopoietic growth factors: at least 14 days after the last dose of a long-acting growth factor (e.g. Neulasta) or 7 days for short-acting growth factor; for agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair
  * Biologic (anti-neoplastic agent): at least 7 days after the last dose of a biologic agent; for agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair
  * Immunotherapy: at least 42 days after the completion of any type of immunotherapy, e.g. tumor vaccines
  * Monoclonal antibodies: at least 3 half-lives of the antibody after the last dose of a monoclonal antibody
  * Radiation therapy (XRT): at least 14 days after local palliative XRT (small port); at least 42 days must have elapsed if other substantial bone marrow (BM) radiation; patients with prior total body irradiation (TBI), craniospinal XRT and/or >= 50% radiation of the pelvis are not eligible
  * Stem cell infusion without TBI: no evidence of active graft vs. host disease and at least 84 days must have elapsed after transplant or stem cell infusion
* PARP inhibitor exposure:

  * Part A: Patients who have received prior therapy with a PARP inhibitor, with the exception of BMN 673, are eligible; however, patients who have progressed on a PARP inhibitor and temozolomide regimen are not eligible
  * Part B: Patients who have previously been exposed to a PARP inhibitor are not eligible
* For patients with solid tumors without known bone marrow involvement: peripheral absolute neutrophil count (ANC) >= 1000/mm^3
* For patients with solid tumors without known bone marrow involvement: platelet count >= 100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
* For patients with solid tumors without known bone marrow involvement: hemoglobin >= 8.0 g/dL (may receive red blood cell [RBC] transfusions)
* All patients enrolled on Part A of the study must be evaluable for hematologic toxicity
* Patients on Part B of the study with known bone marrow metastatic disease will be eligible for the study provided they meet the blood counts (may receive transfusions provided they are not known to be refractory to red cell or platelet transfusions); these patients will not be evaluable for hematologic toxicity
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 ml/min/1.73 m^2 or a maximum serum creatinine (mg/dL) based on age/gender as follows:

  * 1 to < 2 years: 0.6
  * 2 to < 6 years: 0.8
  * 6 to < 10 years: 1
  * 10 to < 13 years: 1.2
  * 13 to < 16 years: 1.5 for males, 1.4 for females
  * >= 16 years: 1.7 for males, 1.4 for females
* Patients on Part A and Part B: bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age
* Patients on Part A and Part B: serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 110 U/L; for the purpose of this study, the ULN for SGPT is 45 U/L
* Patients on Part A and Part B: serum albumin >= 2 g/dL
* All patients and/or their parents or legally authorized representatives must sign a written informed consent; assent, when appropriate, will be obtained according to institutional guidelines
* For patients enrolling on Part B: tissue blocks or slides must be sent; if tissue blocks or slides are unavailable, the Study Chair must be notified prior to enrollment

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study; pregnancy tests must be obtained in girls who are post-menarchal; males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method
* Patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment are not eligible
* Patients who are currently receiving another investigational drug are not eligible
* Patients who are currently receiving other anti-cancer agents are not eligible (except leukemia patients receiving hydroxyurea, which may be continued until 24 hours prior to start of protocol therapy); patients with acute lymphoblastic leukemia may receive intrathecal therapy
* Patients who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease post bone marrow transplant are not eligible for this trial
* Patients must be able to swallow capsules whole
* Patients who have an uncontrolled infection are not eligible
* Patients who have received a prior solid organ transplantation are not eligible
* Patients with prior TBI, craniospinal XRT and/or those with >= 50% radiation of the pelvis are not eligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible
* Patients with known hypersensitivity to temozolomide or dacarbazine are not eligible
* Phase 1 (Part A): patients who have progressed on a PARP inhibitor and temozolomide regimen are not eligible
* Phase 2 (Part B): patients who have previously been exposed to a PARP inhibitor are not eligible
* Phase 1 (Part A): patients with known bone marrow involvement are not eligible

Ages: 13 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2014-05-16 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric S Schafer, Principal Investigator — COG Phase I Consortium
Locations (22):
- United States (22):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Schafer ES, Rau RE, Berg SL, Liu X, Minard CG, Bishop AJR, Romero JC, Hicks MJ, Nelson MD Jr, Voss S, Reid JM, Fox E, Weigel BJ, Blaney SM. Phase 1/2 trial of talazoparib in combination with temozolomide in children and adolescents with refractory/recurrent solid tumors including Ewing sarcoma: A Children's Oncology Group Phase 1 Consortium study (ADVL1411). Pediatr Blood Cancer. 2020 Feb;67(2):e28073. doi: 10.1002/pbc.28073. Epub 2019 Nov 14. PMID 31724813

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients receive talazoparib PO QD or BID on days 1-6 and temozolomide PO QD on days 2-6. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
Groups:
- 400 mcg/m²/Dose BMN 673 QD+20mg/m²/Dose TEM,Max 800 mcg/Day; 400 mcg/m²/Dose BMN 673 BID+20mg/m²/Dose TEM,Max 800 mcg/Day; 600 mcg/m²/Dose BMN 673 BID+20mg/m²/Dose TEM,Max 1000 mcg/Day; 600 mcg/m²/Dose BMN 673 BID+30mg/m²/Dose TEM, Max 1000 mcg/Day; 600 mcg/m²/Dose BMN 673 BID+40mg/m²/Dose TEM, Max 1000 mcg/Day; 600 mcg/m²/doseBMN 673 BID+55mg/m²/Dose TEM, Max 1000 mcg/Day: Phase 1: Part A
  Part A1: Patients with relapsed or refractory solid tumors and CNS tumors
  Part A2: Patients with relapsed or refractory Ewing sarcoma or Peripheral PNET
- 600 mcg/m²/Dose BMN 673 BID+30mg/m²/Dose TEM,Max 1000 mcg/Day: Phase 2: Part B
  Part B: Patients with relapsed or refractory Ewing sarcoma or Peripheral PNET (Phase 2)
Period: Overall Study
Arm/Group | 400 mcg/m²/Dose BMN 673 QD+20mg/m²/Dose TEM,Max 800 mcg/Day | 400 mcg/m²/Dose BMN 673 BID+20mg/m²/Dose TEM,Max 800 mcg/Day | 600 mcg/m²/Dose BMN 673 BID+20mg/m²/Dose TEM,Max 1000 mcg/Day | 600 mcg/m²/Dose BMN 673 BID+30mg/m²/Dose TEM, Max 1000 mcg/Day | 600 mcg/m²/Dose BMN 673 BID+40mg/m²/Dose TEM, Max 1000 mcg/Day | 600 mcg/m²/doseBMN 673 BID+55mg/m²/Dose TEM, Max 1000 mcg/Day | 600 mcg/m²/Dose BMN 673 BID+30mg/m²/Dose TEM,Max 1000 mcg/Day
Started | 3 | 3 | 3 | 13 | 6 | 3 | 9
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 3 | 13 | 6 | 3 | 9
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 2 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 3 | 3 | 3 | 8 | 4 | 1 | 9
Not completed — Physician Decision | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 400 mcg/m²/Dose BMN 673 QD+20mg/m²/Dose TEM,Max 800 mcg/Day | 400 mcg/m²/Dose BMN 673 BID+20mg/m²/Dose TEM,Max 800 mcg/Day | 600 mcg/m²/Dose BMN 673 BID+20mg/m²/Dose TEM,Max 1000 mcg/Day | 600 mcg/m²/Dose BMN 673 BID+30mg/m²/Dose TEM, Max 1000 mcg/Day | 600 mcg/m²/Dose BMN 673 BID+40mg/m²/Dose TEM, Max 1000 mcg/Day | 600 mcg/m²/doseBMN 673 BID+55mg/m²/Dose TEM, Max 1000 mcg/Day | 600 mcg/m²/Dose BMN 673 BID+30mg/m²/Dose TEM,Max 1000 mcg/Day | Total
Number analyzed (Participants) | 3 | 3 | 3 | 13 | 6 | 3 | 9 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 | 3 | 12 | 5 | 3 | 3 | 30
  Between 18 and 65 years | 1 | 1 | 0 | 1 | 1 | 0 | 6 | 10
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: Years] | 18 [16 to 19] | 16 [7 to 19] | 14 [13 to 14] | 13 [5 to 19] | 13.5 [4 to 20] | 12 [6 to 15] | 22 [16 to 25] | 15.5 [4 to 25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 3 | 4 | 2 | 4 | 16
  Male | 2 | 2 | 2 | 10 | 2 | 1 | 5 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 2 | 0 | 0 | 1 | 6
  Not Hispanic or Latino | 3 | 1 | 2 | 11 | 6 | 2 | 7 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 4
  White | 2 | 3 | 2 | 7 | 5 | 2 | 8 | 29
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 3 | 0 | 1 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Dose Limiting Toxicities to Determine the Maximum Tolerated Dose of Temozolomide and Talazoparib Combination Therapy
Description: The Maximum Tolerated Dose (MTD) reflects the highest dose of Talazoparib (BMN 673) when combined with a dose of temozolomide that did not cause a Grade 3 or higher toxicity in children with refractory or recurrent solid tumors.
Time Frame: 28 days
Population: Patients with toxicity grade 3 or above.
Measure: Count of Participants; unit: Participants
Groups:
- 600 mcg/m²/Dose BMN 673 BID+30 mg/m²/Dose TEM,Max 1000 mcg/Day: Part PK
Arm/Group | 400 mcg/m²/Dose BMN 673 QD+20mg/m²/Dose TEM,Max 800 mcg/Day | 400 mcg/m²/Dose BMN 673 BID+20mg/m²/Dose TEM,Max 800 mcg/Day | 600 mcg/m²/Dose BMN 673 BID+20mg/m²/Dose TEM,Max 1000 mcg/Day | 600 mcg/m²/Dose BMN 673 BID+30mg/m²/Dose TEM, Max 1000 mcg/Day | 600 mcg/m²/Dose BMN 673 BID+40mg/m²/Dose TEM, Max 1000 mcg/Day | 600 mcg/m²/doseBMN 673 BID+55mg/m²/Dose TEM, Max 1000 mcg/Day | 600 mcg/m²/Dose BMN 673 BID+30 mg/m²/Dose TEM,Max 1000 mcg/Day
Number analyzed (Participants) | 3 | 3 | 3 | 7 | 6 | 3 | 6
Participants | 0 | 0 | 1 | 2 | 2 | 2 | 0
Statistical Analysis 1: Comparison: 400 mcg/m²/Dose BMN 673 QD+20mg/m²/Dose TEM,Max 800 mcg/Day vs 400 mcg/m²/Dose BMN 673 BID+20mg/m²/Dose TEM,Max 800 mcg/Day vs 600 mcg/m²/Dose BMN 673 BID+20mg/m²/Dose TEM,Max 1000 mcg/Day vs 600 mcg/m²/Dose BMN 673 BID+30mg/m²/Dose TEM, Max 1000 mcg/Day vs 600 mcg/m²/Dose BMN 673 BID+40mg/m²/Dose TEM, Max 1000 mcg/Day vs 600 mcg/m²/doseBMN 673 BID+55mg/m²/Dose TEM, Max 1000 mcg/Day vs 600 mcg/m²/Dose BMN 673 BID+30 mg/m²/Dose TEM,Max 1000 mcg/Day; Test type: Other — Maximum Tolerate Dose Level was determined by the rolling-6 design; Maximum Tolerate Dose Level = 4 — Maximum Tolerate Dose Level is Dose Level 4 (600 mcg/m²/dose +30 mg/m2/dose (BMN 673) BID + 30 mg/m²/dose (TEM), Max 1000 mcg/day). MTD determined by using the Rolling-6 Design

2. Primary Outcome: All Cycle 1 Toxicities >=Grade 3
Description: The number of patients with at least one toxicity (DLT or non-DLT) in cycle 1 that is at least possibly attributable to study agent
Time Frame: Up to 28 days
Population: Patients with toxicity grade 3 or above.
Measure: Count of Participants; unit: Participants
Arm/Group | 400 mcg/m²/Dose BMN 673 QD+20mg/m²/Dose TEM,Max 800 mcg/Day | 400 mcg/m²/Dose BMN 673 BID+20mg/m²/Dose TEM,Max 800 mcg/Day | 600 mcg/m²/Dose BMN 673 BID+20mg/m²/Dose TEM,Max 1000 mcg/Day | 600 mcg/m²/Dose BMN 673 BID+30mg/m²/Dose TEM, Max 1000 mcg/Day | 600 mcg/m²/Dose BMN 673 BID+40mg/m²/Dose TEM, Max 1000 mcg/Day | 600 mcg/m²/doseBMN 673 BID+55mg/m²/Dose TEM, Max 1000 mcg/Day | 600 mcg/m²/Dose BMN 673 BID+30mg/m²/Dose TEM,Max 1000 mcg/Day
Number analyzed (Participants) | 3 | 3 | 3 | 13 | 6 | 3 | 9
Participants | 0 | 0 | 2 | 7 | 5 | 3 | 5

3. Primary Outcome: T Max of Talazoparib
Description: Median with minimum and maximum for the time at which the maximum (peak) serum concentration occurs.
Time Frame: Cycle 1 Day 1 pre-dose, and 1, 2, 4, 8 and 24 hours after the first talazoparib dose.
Population: Pharmacokinetic (PK) studies were completed for all but 3 patients in Phase 1. PK analysis was performed regardless of dose level as pre-specified in the protocol. PK was not performed in Phase 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Treatment (Talazoparib, Temozolomide): Phase 1
Number analyzed (Participants) | 28
Hours | 2 [1 to 24]

4. Primary Outcome: C Max of Talazoparib
Description: Median with minimum and maximum for the time at which the maximum (peak) serum concentration occurs.
Time Frame: Cycle 1 Day 1 pre-dose, and 1, 2, 4, 8 and 24 hours after the first talazoparib dose.
Population: as for outcome 3
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Treatment (Talazoparib, Temozolomide): Phase 1
Number analyzed (Participants) | 28
ng/mL | 4670 [708 to 19300]

5. Primary Outcome: AUC of Talazoparib
Description: Median with minimum and maximum for the area under the drug concentration over time curve.
Time Frame: Cycle 1 Day 1 pre-dose, and 1, 2, 4 and 8 hours after the first talazoparib dose
Population: Pharmacokinetic (PK) studies were completed for all but 4 patients in Phase 1. PK analysis was performed regardless of dose level as pre-specified in the protocol. PK was not performed in Phase 2
Measure: Median (Full Range); unit: h•µg/L
Arm/Group | Treatment (Talazoparib, Temozolomide): Phase 1
Number analyzed (Participants) | 27
h•µg/L | 17.55 [2.15 to 63.14]

6. Primary Outcome: Accumulation Half-life of Talazoparib in Combination With Temozolomide.
Description: Median with minimum and maximum for the time required for the serum concentration to fall to 50% of its starting dose.
Time Frame: Cycle 1 Day 1 pre-dose, and 1, 2, 4 and 8 hours after the first talazoparib dose. Day 5 or 6 pre-dose, and 1, 2, 4 and 8 hours after the talazoparib dose
Population: as for outcome 5
Measure: Median (Full Range); unit: Hours
Arm/Group | Treatment (Talazoparib, Temozolomide): Phase 1
Number analyzed (Participants) | 27
Hours | 46.8 [18.20 to 253.27]

7. Primary Outcome: T Max of Talazoparib in Combination With Temozolomide
Description: Median with minimum and maximum for the time at which the maximum (peak) serum concentration occurs.
Time Frame: Cycle 1 Day 5 or 6 pre-dose, and 1, 2, 4 and 8 hours after the talazoparib dose
Population: as for outcome 3
Measure: Median (Full Range); unit: Hours
Arm/Group | Treatment (Talazoparib, Temozolomide): Phase 1
Number analyzed (Participants) | 28
Hours | 1.04 [1 to 8]

8. Primary Outcome: C Max of Talazoparib in Combination With Temozolomide
Description: Median with minimum and maximum for the time at which the maximum (peak) serum concentration occurs.
Time Frame: Cycle 1 Day 5 or 6 pre-dose, and 1, 2, 4 and 8 hours after the talazoparib dose
Population: as for outcome 3
Measure: Median (Full Range); unit: pg/ml
Arm/Group | Treatment (Talazoparib, Temozolomide): Phase 1
Number analyzed (Participants) | 28
pg/ml | 16450 [7070 to 56300]

9. Primary Outcome: AUC of Talazoparib in Combination With Temozolomide
Description: Median with minimum and maximum area under the drug concentration over time curve
Time Frame: Cycle 1 Day 5 or 6 pre-dose, and 1, 2, 4 and 8 hours after the talazoparib dose
Population: as for outcome 3
Measure: Median (Full Range); unit: h•µg/L
Arm/Group | Treatment (Talazoparib, Temozolomide): Phase 1
Number analyzed (Participants) | 28
h•µg/L | 82.08 [41.92 to 226.70]

10. Primary Outcome: AUC of Talazoparib in Combination With Temozolomide
Description: Median with minimum and maximum area under the drug concentration over time curve
Time Frame: Cycle 1 Day 5 or 6 pre-dose, and 1, 2, 4 and 8 hours after the talazoparib dose
Population: as for outcome 3
Measure: Median (Full Range); unit: h•µg/L
Arm/Group | Treatment (Talazoparib, Temozolomide): Phase 1
Number analyzed (Participants) | 28
h•µg/L | 173.08 [83.61 to 456.28]

11. Primary Outcome: Clearance of Talazoparib in Combination With Temozolomide
Description: Median with minimum and maximum for the rate of elimination of the drug.
Time Frame: Cycle 1 Day 5 or 6 pre-dose, and 1, 2, 4 and 8 hours after the talazoparib dose
Population: as for outcome 3
Measure: Median (Full Range); unit: L/hr/m²
Arm/Group | Treatment (Talazoparib, Temozolomide): Phase 1
Number analyzed (Participants) | 28
L/hr/m² | 3.08 [1.34 to 6.19]

12. Primary Outcome: Accumulation Ratio of Talazoparib in Combination With Temozolomide
Description: Median with minimum and maximum of the accumulation ratio.
Time Frame: as for outcome 6
Population: as for outcome 5
Measure: Median (Full Range); unit: Ratio
Arm/Group | Treatment (Talazoparib, Temozolomide): Phase 1
Number analyzed (Participants) | 27
Ratio | 3.34 [1.67 to 15.73]

13. Primary Outcome: Half-life of Temozolomide in Combination With Talazoparib
Description: Median with minimum and maximum for the time required for the serum concentration to fall to 50% of its starting dose.
Time Frame: Cycle 1 Day 5 or 6 pre-dose, and 1, 2, 4 and 8 hours after the temozolomide dose
Population: Pharmacokinetic (PK) studies were completed for all but 1 patient in Phase 1. PK analysis was performed regardless of dose level as pre-specified in the protocol. PK was not performed in Phase 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Treatment (Talazoparib, Temozolomide): Phase 1
Number analyzed (Participants) | 30
Hours | 1.74 [1.33 to 4.92]

14. Primary Outcome: T Max of Temozolomide in Combination With Talazoparib
Description: Median with minimum and maximum for the time at which the maximum (peak) serum concentration occurs.
Time Frame: Cycle 1 Day 5 or 6 pre-dose, and 1, 2, 4 and 8 hours after the temozolomide dose
Population: as for outcome 13
Measure: Median (Full Range); unit: Hours
Arm/Group | Treatment (Talazoparib, Temozolomide): Phase 1
Number analyzed (Participants) | 30
Hours | 1.03 [1 to 4]

15. Primary Outcome: C Max of Temozolomide in Combination With Talazoparib
Description: Median with minimum and maximum for the maximum (peak) serum concentration.
Time Frame: Cycle 1 Day 5 or 6 pre-dose, and 1, 2, 4 and 8 hours after the temozolomide dose
Population: as for outcome 13
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Treatment (Talazoparib, Temozolomide): Phase 1
Number analyzed (Participants) | 30
ng/mL | 1234.1 [346.56 to 6593.17]

16. Primary Outcome: AUC of Temozolomide in Combination With Talazoparib
Description: Median with minimum and maximum for the area under the drug concentration over time curve.
Time Frame: Cycle 1 Day 5 or 6 pre-dose, and 1, 2, 4 and 8 hours after the temozolomide dose.
Population: as for outcome 13
Measure: Median (Full Range); unit: h•µg/L
Arm/Group | Treatment (Talazoparib, Temozolomide): Phase 1
Number analyzed (Participants) | 30
h•µg/L | 4352.16 [1174.08 to 21653.96]

17. Primary Outcome: Clearance of Temozolomide in Combination With Talazoparib
Description: Median with minimum and maximum for the rate of elimination of the drug.
Time Frame: Cycle 1 Day 5 or 6 pre-dose, and 1, 2, 4 and 8 hours after the temozolomide dose
Population: as for outcome 13
Measure: Median (Full Range); unit: L/hr/m²
Arm/Group | Treatment (Talazoparib, Temozolomide): Phase 1
Number analyzed (Participants) | 30
L/hr/m² | 6.49 [2.59 to 30.08]

18. Primary Outcome: Number of Ewing/Peripheral PNET Participants in Phase 2 With Complete Response (CR) or Partial Response (PR)
Description: Frequency of Ewing sarcoma and peripheral PNET participants with Complete Response (CR) or Partial Response (PR) per the Response Evaluation Criteria In Solid Tumors (RECIST)
Time Frame: Up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Talazoparib, Temozolomide): Phase 2
Number analyzed (Participants) | 9
Participants | 0

19. Secondary Outcome: Number of Solid Tumor Patients With Complete Response (CR) or Partial Response (PR)
Description: Frequency of solid tumor participants with Complete Response (CR) or Partial Response (PR) per the Response Evaluation Criteria In Solid Tumors (RECIST)
Time Frame: Up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Talazoparib, Temozolomide): Phase 1
Number analyzed (Participants) | 31
Participants | 1

ADVERSE EVENTS:
Time Frame: Up to 24 months
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Arm/Group | 400 mcg/m²/Dose BMN 673 QD+20mg/m²/Dose TEM,Max 800 mcg/Day | 400 mcg/m²/Dose BMN 673 BID+20mg/m²/Dose TEM,Max 800 mcg/Day | 600 mcg/m²/Dose BMN 673 BID+20mg/m²/Dose TEM,Max 1000 mcg/Day | 600 mcg/m²/Dose BMN 673 BID+30mg/m²/Dose TEM, Max 1000 mcg/Day | 600 mcg/m²/Dose BMN 673 BID+40mg/m²/Dose TEM, Max 1000 mcg/Day | 600 mcg/m²/doseBMN 673 BID+55mg/m²/Dose TEM, Max 1000 mcg/Day | 600 mcg/m²/Dose BMN 673 BID+30mg/m²/Dose TEM,Max 1000 mcg/Day
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 2/13 | 1/6 | 0/3 | 0/9
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 2/3 | 11/13 | 6/6 | 3/3 | 8/9
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 13/13 | 6/6 | 3/3 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 400 mcg/m²/Dose BMN 673 QD+20mg/m²/Dose TEM,Max 800 mcg/Day (N=3) | 400 mcg/m²/Dose BMN 673 BID+20mg/m²/Dose TEM,Max 800 mcg/Day (N=3) | 600 mcg/m²/Dose BMN 673 BID+20mg/m²/Dose TEM,Max 1000 mcg/Day (N=3) | 600 mcg/m²/Dose BMN 673 BID+30mg/m²/Dose TEM, Max 1000 mcg/Day (N=13) | 600 mcg/m²/Dose BMN 673 BID+40mg/m²/Dose TEM, Max 1000 mcg/Day (N=6) | 600 mcg/m²/doseBMN 673 BID+55mg/m²/Dose TEM, Max 1000 mcg/Day (N=3) | 600 mcg/m²/Dose BMN 673 BID+30mg/m²/Dose TEM,Max 1000 mcg/Day (N=9)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 1 | 2 | 5
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Catheter related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Dysphasia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Edema face (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Fever (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
GGT increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypersomnia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Irregular menstruation (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 2 | 0 | 4 | 2 | 2 | 6
Lymphocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, PROGRESSIVE DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, PROGRESSIVE DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nervous system disorders - Other, HYPOTONIC (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nervous system disorders - Other, PARALYSIS (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 8 | 5 | 3 | 5
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Oculomotor nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Optic nerve disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Periorbital infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 4 | 3 | 2 | 5
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, VOCAL CORD PARALYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Typhlitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Weight loss (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell decreased (Investigations) | 0 | 0 | 0 | 3 | 2 | 2 | 5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 400 mcg/m²/Dose BMN 673 QD+20mg/m²/Dose TEM,Max 800 mcg/Day (N=3) | 400 mcg/m²/Dose BMN 673 BID+20mg/m²/Dose TEM,Max 800 mcg/Day (N=3) | 600 mcg/m²/Dose BMN 673 BID+20mg/m²/Dose TEM,Max 1000 mcg/Day (N=3) | 600 mcg/m²/Dose BMN 673 BID+30mg/m²/Dose TEM, Max 1000 mcg/Day (N=13) | 600 mcg/m²/Dose BMN 673 BID+40mg/m²/Dose TEM, Max 1000 mcg/Day (N=6) | 600 mcg/m²/doseBMN 673 BID+55mg/m²/Dose TEM, Max 1000 mcg/Day (N=3) | 600 mcg/m²/Dose BMN 673 BID+30mg/m²/Dose TEM,Max 1000 mcg/Day (N=9)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 2 | 2 | 2
Abducens nerve disorder (Nervous system disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 3 | 4 | 1 | 3
Alkaline phosphatase increased (Investigations) | 1 | 1 | 1 | 2 | 1 | 1 | 7
Allergic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 6 | 2 | 1 | 3
Anemia (Blood and lymphatic system disorders) | 2 | 2 | 2 | 12 | 6 | 3 | 8
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 7 | 1 | 2 | 3
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 4 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 1 | 2 | 2 | 1 | 5
Ataxia (Nervous system disorders) | 0 | 1 | 1 | 3 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 3 | 3 | 2 | 3
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 2 | 1 | 0 | 3
Blurred vision (Eye disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Brachial plexopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2 | 1 | 1 | 0
Burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 1 | 0 | 0
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac disorders - Other, HEART MURMUR (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac disorders - Other, MURMUR LUSB (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac disorders - Other, NON RESTRICTIVE CARDIOMYOPATHY (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Cholesterol high (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Concentration impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 5 | 4 | 2 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 3 | 3 | 1 | 2
Creatinine increased (Investigations) | 1 | 0 | 1 | 4 | 3 | 2 | 3
Cushingoid (Endocrine disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 1 | 5 | 2 | 1 | 3
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 2 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0
Dysphasia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 2
Ear and labyrinth disorders - Other, DECREASED HEARING (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear and labyrinth disorders - Other, HEARING LOSS (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Edema limbs (General disorders) | 1 | 0 | 0 | 3 | 3 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Endocrine disorders - Other, PANHYPOPITUITARISM (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 1 | 0 | 1
Esophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye disorders - Other, DOUBLE VISION (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Eye disorders - Other, LEFT ORBITAL RECONSTRUCTION (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye disorders - Other, SPOTS IN VISUAL FIELD (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye disorders - Other, VISION IMPAIRMENT (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Facial nerve disorder (Nervous system disorders) | 0 | 1 | 1 | 5 | 1 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 1 | 0 | 10 | 5 | 3 | 6
Fecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fever (General disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 1 | 0 | 2 | 1 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 1 | 0 | 1
Gastrointestinal disorders - Other, GINGIVAL BLEEDING (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal disorders - Other, OROPHARYNGEAL ERYTHEMA (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal disorders - Other, VOMITING WITH BLOOD STREAKS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 2 | 0 | 0
Glossopharyngeal nerve disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hallucinations (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 1 | 1 | 3 | 0 | 3 | 5
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Hematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hemoglobin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hemoglobinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 1 | 2 | 5 | 2 | 0 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 3 | 0 | 0 | 5
Hypernatremia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2 | 0 | 0 | 2
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 2 | 2 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 5 | 3 | 2 | 4
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 1 | 2 | 3
Hypoglossal nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 1 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2 | 0 | 2 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1 | 2 | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 4 | 2 | 0 | 2
Hypotension (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 2
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
IVth nerve disorder (Nervous system disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0
Infections and infestations - Other, HHV6 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infections and infestations - Other, SHINGLES ZOSTER (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infections and infestations - Other, THRUSH (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infections and infestations - Other, URI (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injury, poisoning and procedural complications - Other, EAR CUT (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injury, poisoning and procedural complications - Other, LEG LACERATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injury, poisoning and procedural complications - Other, SCRATCHES (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 1 | 0 | 2 | 0 | 1
Intraoperative neurological injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Investigations - Other, ALK PHOS DECREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Investigations - Other, ALT DECREASED (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, ANION GAP INCREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Investigations - Other, AST DECREASED (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, BICARBONATE DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Investigations - Other, BICARBONATE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Investigations - Other, BICARBONATE LOW (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Investigations - Other, BICARBONATE SERUM LOW (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, BUN DECREASED (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Investigations - Other, CHLORIDE INCREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Investigations - Other, ELEVATED BUN (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, ELEVATED LDH (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, HARD STOOL (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Investigations - Other, HCT INCREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Investigations - Other, HIGH PLATELET COUNT (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Investigations - Other, HYPOCHLOREMIA (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Investigations - Other, INCREASED WBC L (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Investigations - Other, LOW BICARBONATE (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Investigations - Other, MONOCYTE COUNT INCREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Investigations - Other, NEUTROPHIL COUNT INCREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Investigations - Other, PLATELETS INCREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Irritability (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0
Lip infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphedema (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 2 | 2 | 10 | 4 | 1 | 4
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Metabolism and nutrition disorders - Other, CHLORIDE LEVEL (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 1
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0
Musculoskeletal and connective tissue disorder - Other, L WRIST CONTRACTURE (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, LARGE OCCIPITAL SKULL DEFECT (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal and connective tissue disorder - Other, LEG CRAMPS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, LEG SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 1 | 3 | 6 | 4 | 2 | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 2
Nervous system disorders - Other, DIFFICULTIES WITH BALANCE (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nervous system disorders - Other, LEFT HEMIPLEGIA (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 2 | 1 | 7 | 3 | 0 | 5
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 4
Nystagmus (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oculomotor nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 3 | 3 | 2 | 5
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Papulopustular rash (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paresthesia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Penile pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 2 | 1 | 1 | 9 | 4 | 2 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 1
Precocious puberty (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Psychiatric disorders - Other, HX OF ADHD (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyramidal tract syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0
Recurrent laryngeal nerve palsy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal and urinary disorders - Other, BLADDER PAIN (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal and urinary disorders - Other, GLUCOSE IN URINE (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, OBSTRUCTIVE SLEEP APNEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, REQUIRES TRACH WITH FLOW OVERNIGHT (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, RETRACTIONS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, RHINORRHEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, TACHYPNEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 1 | 5 | 2 | 3 | 3
Skin and subcutaneous tissue disorders - Other, ABRASION ON LEG (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin and subcutaneous tissue disorders - Other, LEFT LOWER LEG ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, MOM NOTICED DARK VEINS ON BACK (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, PEELING LEFT HEEL (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other, PEELING SKIN ON HEEL AREA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other, PEELING SKIN, FINGERTIPS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, POISON IVY RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, RASH (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, RED HANDS AND CHEEKS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, RIGHT UPPER HEAD AND RIGHT POSTERIOR HEAD LESION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, SKIN LESIONS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, TENDERNESS OVER SPINE (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 0 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2 | 1 | 1 | 0
Spasticity (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 0 | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urine discoloration (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 5 | 4 | 3 | 3
Weight gain (Investigations) | 0 | 0 | 0 | 1 | 2 | 0 | 0
Weight loss (Investigations) | 1 | 0 | 0 | 2 | 1 | 2 | 1
White blood cell decreased (Investigations) | 1 | 2 | 2 | 10 | 5 | 3 | 7
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-23): https://cdn.clinicaltrials.gov/large-docs/77/NCT02116777/Prot_SAP_001.pdf